CLINICAL TRIAL: NCT00829101
Title: Articulatory and Phonological Competence at 3 and 5 Years of Age in Children With Unilateral Cleft Lip and Palate Who Have Undergone Different Methods of Primary Palatal Surgery
Brief Title: Articulation and Phonology in Children With Unilateral Cleft Lip and Palate
Acronym: APCLP
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Karolinska Institutet (Other); Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: D-nr: 548/2008
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Cleft Palate; Cleft Lip
Keywords: unilateral cleft lip and palate; primary palatal surgery; articulation; phonology; one stage palatal repair; two stage palatal repair
MeSH Terms: conditions — Cleft Palate; Cleft Lip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1 One-stage repair: A consecutive group of children born with unilateral cleft lip and palate from the south region of Sweden, in all 10 children, who have had a primary palatal surgery at 12 months of age.
- 2 Two-stage repair, early closure: A consecutive group of children born with unilateral cleft lip and palate from the western region of Sweden, in all 10 children, who have had a two-stage palatal surgery, with soft palate closure at 4-6 months and repair of the hard palate at 12 months of age.
- 3 Two-stage repair, delayed closure: A consecutive group of children born with unilateral cleft lip and palate from the western region of Sweden, in all 10 children, who have have had a two-stage palatal surgery, with soft palate closure at 4-6 months and repair of the hard palate at 36 months of age.

SUMMARY:
The purpose of the study is to assess if there are any differences in the articulatory and phonological competence in pre-school children with unilateral cleft lip and palate (UCLP) who are treated with different surgical methods of palatal repair.

DETAILED DESCRIPTION:
A cleft palate may influence important functions such as eating, function of the ear/hearing, speech, occlusion, and in addition social skills and acceptability related to appearance. Surgical treatment is aiming to minimize the impact of the cleft on these functions. Nevertheless there is often a need of orthodontic treatment, and if the palate is involved, speech therapy and speech improving secondary surgery. The incidence of otitis media with effusion, and related hearing problems, is high among the children. The outcome is affected by type of cleft as well as surgical method, although not yet fully clarified. Some consider the growth of the mid-face to be better if primary surgery of the hard palate is delayed, while speech development is considered to benefit from primary palate surgery performed as early as possible. Yet we don´t know which surgical method is the best. In most parts of the world and at three of six treatment centers in Sweden the palate is closed in one stage between 12 and 18 months of age. At the three other Swedish centers the cleft in the soft palate is closed at 4-6 months, and the cleft in the hard palate is repaired at 2-3 years of age.

Video-recordings of the children at 3 and 5 years of age will be used for evaluation. The speech material at 3 years of age consists of spontaneous speech and word naming. At 5 years sentence repetition and a re-telling task is added. Blindly transcription of the material after randomization, according to the transcription used for cleft palate speech in Sweden based on the IPA and ExtIPA conventions will be performed. About 30% of the material, randomly selected, will be re-transcribed and about 30% will be transcribed by an additional listener independently, for calculation of reliability. The results will be compared between groups regarding articulatory deviancies and phonological processes, and will be statistically analyzed. Impact of ear problems, hearing and speech therapy will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* born with unilateral cleft lip and palate
* native Swedish speaking

Exclusion Criteria:

* known syndromes and/or additional malformations

Ages: 3 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children from the south or western region of Sweden born with unilateral cleft lip and palate.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Percent correct consonants | 3 and 5 years of age

SECONDARY OUTCOMES:
Phonological simplification processes | 3 and 5 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Henry Svensson, Professor, Head, Study Director — Department of Plastic and reconstructive Surgery, Skåne University Hospital, Sweden
Locations (1):
- Department of Logopedics, Skåne University Hospital Malmö, Malmo, Region Skane, Sweden

REFERENCES:
- [Background] Farzaneh F, Lindman R, Becker M, Hansen K, Svensson H. von Langenbeck procedures at 8 months or Wardill at 18 months for primary repair of cleft palate in adult Swedish patients with unilateral complete cleft lip and palate: a study of facial growth. Scand J Plast Reconstr Surg Hand Surg. 2008;42(2):67-76. doi: 10.1080/02844310701850512. PMID 18335350
- [Background] Farzaneh F, Becker M, Peterson AM, Svensson H. Speech results in adult Swedish patients born with unilateral complete cleft lip and palate. Scand J Plast Reconstr Surg Hand Surg. 2008;42(1):7-13. doi: 10.1080/02844310701694522. PMID 18188776
- [Background] Friede H. Maxillary growth controversies after two-stage palatal repair with delayed hard palate closure in unilateral cleft lip and palate patients: perspectives from literature and personal experience. Cleft Palate Craniofac J. 2007 Mar;44(2):129-36. doi: 10.1597/06-037.1. PMID 17328651
- [Background] Lohmander A, Persson C. A longitudinal study of speech production in Swedish children with unilateral cleft lip and palate and two-stage palatal repair. Cleft Palate Craniofac J. 2008 Jan;45(1):32-41. doi: 10.1597/06-123.1. PMID 18215097
- [Background] Peterson-Falzone SJ. The relationship between timing of cleft palate surgery and speech outcome: what have we learned, and where do we stand in the 1990s? Semin Orthod. 1996 Sep;2(3):185-91. doi: 10.1016/s1073-8746(96)80013-2. PMID 9161287